CLINICAL TRIAL: NCT07009249
Title: Effects of Dynamic Neuromuscular Stabilization Exercises on Urinary Symptoms and Pelvic Floor Muscle Functions in Women With Stress Urinary Incontinence: A Single-Blind Non-Inferiority Clinical Study
Brief Title: Dynamic Neuromuscular Stabilization Exercises in Women With Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Seda Yakit Yesilyurt, Asst. Prof., Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYY_IEU_5
Record Dates: First submitted 2025-05-21; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Stress Urinary Incontinence (SUI); Dynamic Neuromuscular Stabilization; Pelvic Floor Muscle Training; Urinary Symptoms; Biofeedback Training
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Muscle Training Group (PFMT Group) (Active Comparator): Women aged 18-62 who have stress or stress-dominant mixed urinary incontinence and can read and write in Turkish
  Interventions: Behavioral: Pelvic floor muscle training
- Dynamic Neuromuscular Stabilization Group (DNS Group) (Experimental): Women aged 18-62 who have stress or stress-dominant mixed urinary incontinence and can read and write in Turkish
  Interventions: Behavioral: Dynamic neuromuscular stabilization

INTERVENTIONS:
Behavioral: Pelvic floor muscle training — Women in this group will undergo pelvic floor muscle training (PFMT) using the NeuroTrac MyoPlus 4 PRO EMG biofeedback device. Prior to the training, diaphragmatic breathing will be taught to all participants in this position to facilitate relaxation and prepare for PFMT. During the training, participants will perform pelvic floor muscle contractions while observing the real-time feedback of slow and fast contractions, as well as relaxation phases, on the computer screen connected to the device. Concurrently, the physiotherapist will guide the participants with verbal cues such as "squeeze-lift-release." Participants will be instructed to avoid holding their breath, pulling in their abdomen, straining, contracting the thigh or gluteal muscles, or moving the pelvis during the exercises. The PFMT protocol will follow the principles of motor learning stages to ensure proper skill acquisition.
  Arms: Pelvic Floor Muscle Training Group (PFMT Group)
Behavioral: Dynamic neuromuscular stabilization — Women in this group will be instructed in exercises based on the principles of Dynamic Neuromuscular Stabilization (DNS). Prior to the exercises, intra-abdominal pressure regulation through breathing techniques will be demonstrated. In this study, the Core 360 belt with OhmTrack sensors will be used. Both breathing exercises and DNS exercises will be taught with the belt in place. In a corrected posture, participants will be instructed to gently press the abdominal wall toward the sensors and to maintain expansion of the abdominal wall during both inspiration and expiration, while keeping the spine in a neutral position. The exercise program will begin with a preparatory training phase, which includes fascial mobilizations applied to the feet and hands. DNS exercises will start with the 4.5-month supine developmental position for sagittal stabilization. As the program progresses, exercises will be advanced according to developmental kinesiology positions.
  Arms: Dynamic Neuromuscular Stabilization Group (DNS Group)

SUMMARY:
Stress urinary incontinence (SUI) is defined by the International Continence Society as the complaint of involuntary leakage of urine during physical exertion, including sports activities, or during sneezing or coughing. In continent women, an automatic response-namely, a reflex pelvic floor muscle (PFM) contraction, also known as pre-contraction-occurs either prior to or during physical exertion. Although there is strong evidence supporting the effectiveness of pelvic floor muscle training (PFMT) in the treatment of SUI, there has been a growing interest in exploring alternative exercise-based interventions.

Dynamic Neuromuscular Stabilization (DNS) is a manual and rehabilitative approach developed by Professor Pavel Kolar. It is grounded in the scientific principles of developmental kinesiology and aims to optimize the function of the movement system. Currently, DNS is successfully employed in the rehabilitation of various neurological, musculoskeletal, pediatric, and sports-related injuries. DNS incorporates the subconscious and synergistic activation of the deep core muscles responsible for intra-abdominal pressure (IAP) regulation and spinal stability-namely, the diaphragm, transversus abdominis, multifidus, and pelvic floor muscles-as well as the global musculature.

Considering the potential mechanisms of DNS, we hypothesize that DNS exercises, through IAP regulation directed toward the pelvic cavity and contributing to stabilization, could serve as an effective and innovative approach for women with SUI.

The hypotheses of this study are as follows:

H1.1: DNS is as effective as PFMT in reducing urinary symptoms in women with SUI.

H1.2: DNS is as effective as PFMT in improving PFM function in women with SUI.

ELIGIBILITY:
Inclusion Criteria:

* Female gender,
* Voluntary participation in the study,
* Aged between 18 and 62 years,
* Ability to read and write in Turkish,
* No mental disorders that would impair cooperation or comprehension,
* Complaint of stress urinary incontinence (SUI) or stress-predominant mixed urinary incontinence.

Exclusion Criteria:

* Prior history of pelvic floor muscle training,
* Presence of any neurological disorder,
* Pelvic organ prolapse stage II or higher,
* Presence of fecal incontinence,
* Pregnancy,
* Lower extremity conditions that may affect pelvic alignment (e.g., leg length discrepancy, total hip arthroplasty),
* Active lower urinary tract infection,
* Presence of respiratory disorders such as chronic obstructive pulmonary disease or asthma,
* History of hysterectomy.

Ages: 18 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change of Pelvic Floor Pre-contraction during valsalva | From enrollment to the end of treatment at 8 weeks
  Pre-contraction of PFM during valsalva will be evaluated with NeuroTract Myoplus 4 PRO EMG device.The assessment will be conducted as described in previous studies. Participants will be instructed as follows: "Take a deep breath in, pinch your nose with your thumb and index finger, and close your mouth. Now try to exhale against the closed airway." The reflex activity of the pelvic floor muscles will be recorded in microvolts (μV) over a 2-second interval.

SECONDARY OUTCOMES:
Pelvic floor muscle strength (Vaginal palpation) | From enrollment to the end of treatment at 8 week
  Vaginal palpation method will be used to measure pelvic floor muscle strength. The Modified Oxford Scale will be used in the assessment.(0= no contraction; 1= very weak; 2= weak; 3= moderate (with lifting); 4= good (with lifting); 5= strong (with lifting))
Resting EMG activity | From enrollment to the end of treatment at 8 weeks
  Resting tone of PFM will be evaluated with NeuroTract Myoplus 4 PRO EMG device.Resting tone is defined as vaginal resting activity, and in order to measure resting EMG electrical activity, women will be asked to remain as still as possible, not to perform voluntary PFM contraction or straining, and to maintain their most comfortable positions. After this condition is achieved, the numerical equivalent of the electrical activity occurring in the EMG probe on the monitor will be recorded as resting activity in terms of (μV).
Maximum voluntary contraction | From enrollment to the end of treatment at 8 weeks
  Maximum voluntary contraction of PFM will be evaluated with NeuroTract Myoplus 4 PRO EMG device. After recording the resting EMG activity of the pelvic floor muscles, women will be asked to perform maximum voluntary contraction. Maximum voluntary contraction force (microvolts (μV)) will be automatically recorded by the device after three measurements.
Change in Urinary Incontinence Severity | From enrollment to the end of treatment at 8 weeks
  The severity of urinary incontinence in women will be assessed using the Incontinence Severity Index (ISI). This index consists of two questions. Participants will be asked:
  "How often do you experience urine leakage?" with response options scored as 1 (less than once a month), 2 (a few times a month), 3 (a few times a week), or 4 (every day and/or night); and "How much urine do you usually leak each time?" with options scored as 1 (a few drops), 2 (small splashes), or 3 (more).
  The total score is calculated by multiplying the scores of the two items, resulting in a total score ranging from 1 to 12. Higher scores indicate more severe urinary incontinence.
Change in urinary symptoms and impact on quality of life | From enrollment to the end of treatment at 8 weeks
  Urinary incontinence symptoms and their impact on quality of life will be assessed using the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF). The ICIQ-SF was developed by Avery et al. to evaluate urinary incontinence and its effects on quality of life. The questionnaire has been reported to have high levels of sensitivity, reliability, and validity. Only the first three domains are scored, while the fourth domain provides descriptive information that can help identify the type of urinary incontinence. Each scored domain can be analyzed independently, or the scores of the first three items can be summed to assess the overall impact of urinary incontinence on quality of life. The total score ranges from 0 to 21, with higher scores indicating greater impact on quality of life.
Change of contraction onset time | From enrollment to the end of treatment at 8 weeks
  Contraction of PFM onset time will be evaluated with NeuroTract Myoplus 4 PRO EMG device. Contraction onset time (seconds) will be automatically recorded by the device after three measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yakıt Yeşilyurt, Principal Investigator — Izmir University of Economics
Locations (1):
- Izmir University of Economics, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No